CLINICAL TRIAL: NCT04180319
Title: A Pan-European Multi-Centre Observational Study To Determine The Natural History Of Patients With Alpha-1 Antitrypsin
Brief Title: EARCO REGISTRY. History Of Patients With Alpha-1 Antitrypsin
Acronym: EARCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: European Respiratory Society (Other)
Responsible Party: Sponsor
Other Study IDs: EARCO
Record Dates: First submitted 2019-09-04; First posted 2019-11-27 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-11

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Natural History; Epidemiology; Registry; alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
European Alpha-1 Research Collaboration (EARCO) is a pan-European network committed to promoting clinical research and education in alpha-1 antitrypsin deficiency (AATD). The core project is the pan-European AATD Registry, a collaboration which will offer longitudinal real-world data for patients with AATD. EARCO has a global vision to increase the early diagnosis of alpha-1 antitrypsin deficiency (AATD), understand better the natural history of the disease and ensure optimal access to effective care, placing emphasis on ambitions that serve collective needs of the AATD research community and bringing people with AAT deficiency to the centre of the research environment in a real-world context.

The study population will consist of individuals with diagnosed severe alpha-1 antitrypsin deficiency regardless of the clinical expression and severity.

The study objectives are:

* To generate long-term, high-quality clinical data covering a pan-European population of AATD individuals in all age groups and all stages of disease severity.
* To understand the natural history and prognosis of AATD better with the goal to create and validate prognostic tools to support medical decision making.
* To investigate the effect of augmentation therapy on the progression of emphysema and to examine its impact on clinical and functional outcomes, such as FEV1, quality of life and mortality in a "real-life" population
* To learn more about the course of the disease in patients suffering from severe AATD with genotypes different from Pi*ZZ We expect to collect detailed information from around 1,000 patients from at least 10 countries during the first year, expanding to 3,000 from more than 25 countries over the 5 years of the CRC and continue a long term follow-up.

We expect to collect detailed information from around 1,000 patients from at least 10 countries during the first year, expanding to 3,000 from more than 25 countries over the 5 years of the CRC and continue a long term follow-up. .

DETAILED DESCRIPTION:
EARCO takes advantage of existing AATD registries that have been developed at the national level. Several countries have established registries in which AATD patients are included and followed-up with clinical and biological data collected. However, these registries differ in terms of inclusion criteria, data collected and frequency and extent of follow-up. Within EARCO, we will harmonize the data collection process and assess the quality of the data within a short time frame after the data are generated and entered into the database.

We expect to collect detailed information from around 1,000 patients from at least 10 countries during the first year, expanding to 3,000 from more than 25 countries over the 5 years of the CRC and continue a long term follow-up. .

The study objectives are:

* To generate long-term, high-quality clinical data covering a pan-European population of AATD individuals in all age groups and all stages of disease severity.
* To understand the natural history and prognosis of AATD better with the goal to create and validate prognostic tools to support medical decision making.
* To investigate the effect of augmentation therapy on the progression of emphysema and to examine its impact on clinical and functional outcomes, such as FEV1, quality of life and mortality in a "real-life" population
* To learn more about the course of the disease in patients suffering from severe AATD with genotypes different from Pi*ZZ

Study design:

The EARCO registry is a non-interventional, multi-centre, pan-European, prospective, repetitive, observational cohort study enrolling patients with AATD (as confirmed by serum level and genotyping). Patients will be managed according to their local procedures and policies with no interference from the study team. Patients will give informed consent to participate, and participating investigators will collect data prospectively. The following domains are covered: demographics, proteinase inhibitor genotype and other laboratory analyses, comorbidities, lung function, transient elastography of the liver, exacerbations, quality of life (QoL), chest CT (if applicable), and treatment.

The study protocol was reviewed by the Research Ethics Committee of the Vall d'Hebron University Hospital of Barcelona, Spain, and the study is sponsored by Vall d'Hebron Research Institute, Barcelona, Spain. The study website will be located at www.AATD.eu. The registry was developed according to recommendations on the design, implementation, governance and long-term sustainability of disease registries in the European Union (EU). It is funded as a clinical research collaboration (CRC) under the umbrella of the European Respiratory Society (ERS). Clinical Research Collaborations (CRCs) are pan-European, multi-centre networks of principal investigators aiming to advance science and clinical research within a specific disease area (www.ersnet.org/ers-funding/clinical-research-collaboration.html). The European Alpha-1 Clinical Research Collaboration (EARCO) was established as an ERS CRC with the objective of developing a European AATD Registry and bringing researchers together internationally to promote clinical research, clinical care and education.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Alpha-1 antitrypsin deficiency, defined as

  * AAT serum level < 11 µM (50 mg/dl) and/or
  * proteinase inhibitor genotypes ZZ, SZ, and compound heterozygotes or homozygotes of other rare deficient variants.

Exclusion Criteria:

* Patients unwilling or unable to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of individuals with diagnosed severe alpha-1 antitrypsin deficiency regardless of the clinical expression and severity.
  We expect to collect detailed information from around 1,000 patients from at least 10 countries during the first year, expanding to 3,000 from more than 25 countries over the 5 years of the CRC.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
Evolution of lung function The Natural History Of Patients With Alpha-1 Antitrypsin Deficiency | 5 years
  Annual measurement of forced expiratory volume in the first second (FEV1) in liters
Mortality | 5 years
  Mortality during the duration of the study
Evolution of respiratory specific health related quaility of life | 5 years
  Annual measurements of COPD Assessment Test (CAT) (scale 0 to 40 points)
Evolution of generic health related quaility of life | 5 years
  Annual measurement of EQ-5D

SECONDARY OUTCOMES:
Incidence of liver disease | 5 years
  Alterations in liver enzymes and/or liver imaging tests during follow-up
Evolution of respiratory symptoms | 5 years
  identification of respìratory symptoms during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: MARC MIRAVITLLES, MD-PhD, Principal Investigator — Hospital Vall d'Hebron; Timm Greulich, MD-PhD, Principal Investigator — University Medical Centre Giessen and Marburg, Germany
Locations (1):
- Marc Miravitlles, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miravitlles M, Dirksen A, Ferrarotti I, Koblizek V, Lange P, Mahadeva R, McElvaney NG, Parr D, Piitulainen E, Roche N, Stolk J, Thabut G, Turner A, Vogelmeier C, Stockley RA. European Respiratory Society statement: diagnosis and treatment of pulmonary disease in alpha1-antitrypsin deficiency. Eur Respir J. 2017 Nov 30;50(5):1700610. doi: 10.1183/13993003.00610-2017. Print 2017 Nov. PMID 29191952
- [Background] Miravitlles M, Chorostowska-Wynimko J, Ferrarotti I, McElvaney NG, O'Hara K, Stolk J, Stockley RA, Turner A, Wilkens M, Greulich T; EARCO Clinical Research Collaboration; Members of the EARCO Clinical Research Collaboration. The European Alpha-1 Research Collaboration (EARCO): a new ERS Clinical Research Collaboration to promote research in alpha-1 antitrypsin deficiency. Eur Respir J. 2019 Feb 14;53(2):1900138. doi: 10.1183/13993003.00138-2019. Print 2019 Feb. No abstract available. PMID 30765486
- [Derived] Martin T, Guimaraes C, Esquinas C, Torres-Duran M, Turner AM, Tanash H, Rodriguez-Garcia C, Corsico A, Lopez-Campos JL, Bartosovska E, Staehr Jensen JU, Hernandez-Perez JM, Sucena M, Miravitlles M. Risk of lung disease in the PI*SS genotype of alpha-1 antitrypsin: an EARCO research project. Respir Res. 2024 Jun 26;25(1):260. doi: 10.1186/s12931-024-02879-y. PMID 38926693
- [Derived] Miravitlles M, Turner AM, Torres-Duran M, Tanash H, Rodriguez-Garcia C, Lopez-Campos JL, Chlumsky J, Guimaraes C, Rodriguez-Hermosa JL, Corsico A, Martinez-Gonzalez C, Hernandez-Perez JM, Bustamante A, Parr DG, Casas-Maldonado F, Hecimovic A, Janssens W, Lara B, Barrecheguren M, Gonzalez C, Stolk J, Esquinas C, Clarenbach CF. Clinical and functional characteristics of individuals with alpha-1 antitrypsin deficiency: EARCO international registry. Respir Res. 2022 Dec 16;23(1):352. doi: 10.1186/s12931-022-02275-4. PMID 36527073